CLINICAL TRIAL: NCT05167773
Title: Clinical Study of the Topcon Tonometer TRK-3 to Demonstrate Conformance to ISO 8612, JIS T7312, and ANSI Z80.10-2014 Ophthalmic Instruments - Tonometers
Brief Title: Clinical Study of the Topcon Tonometer TRK-3
Status: Completed | Type: Observational
Sponsor: Topcon Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: THQ-2021-04
Record Dates: First submitted 2021-11-08; First posted 2021-12-22 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Intraocular Pressure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: tonometer — A subject undergoes intraocular pressure measurement with tonometer

SUMMARY:
The study will assess the TRK-3 for conformity to ISO 8612:2009, JIS T7312:2015, and ANSI Z80.10-2014 Ophthalmic Instruments - Tonometers, to the FDA Guidance for Industry and FDA Staff, Tonometer-Premarket Notification [510(k)] Submissions, and the applicable Supplemental Information Sheet.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years of age or older at the time of informed consent
2. Irrespective of sex
3. Irrespective of race or ethnicity
4. Be willing and able to provide written informed consent by subject or legally designated representative prior to any study procedures

Exclusion Criteria:

1. Have only one functional eye
2. Have one eye with poor or eccentric fixation
3. Have corneal scarring or have had corneal surgery, including corneal laser surgery in either eye
4. Have microphthalmos in either eye
5. Have buphthalmos in either eye
6. Be a contact lens wearer (persons wearing soft contact lenses within the past 3 months and/or hard contact lenses within the past 6 months)
7. Have dry eyes (persons who have been diagnosed by a physician and are currently using prescription drugs or routinely using artificial tears)
8. Uncontrollably blink, squint, wink, twitch or squeeze eye(s) - blepharospasm
9. Have nystagmus in either eye
10. Have keratoconus in either eye
11. Have any other corneal or conjunctival pathology or infection in either eye
12. Have central corneal thickness is less than 500μm or more than 600μm
13. Be allergic to eye drop anesthetics
14. Be allergic to sodium fluorescein

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing routine eye exam at eye care clinic
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
fluid pressure inside the eye (intraocular pressure) measured in millimeters of mercury (mm Hg) | 1 day
  Intraocular Pressure (IOP) measurements acquired with the study tonometer are compared to the reference tonometer IOP measurements to demonstrate that they meet the requirement specified in the tonometer standards (ISO 8612:2009, JIS T7312:2015 and ANSI Z80.10-2014)

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Kato Eye Clinic, Tokyo
  - Seiyo Clinic, Tokyo

IPD SHARING:
Plan to Share IPD: No